CLINICAL TRIAL: NCT04018196
Title: Effects of Motor Imagery on Motor Learning and Motor Retention in Octogenarian "IMAge-8".
Brief Title: Effects of Motor Imagery on Motor Learning and Motor Retention in Octogenarian.
Acronym: IMAge-8
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of inclusions
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18CH128; 2018-A02365-50 (Other: ANSM)
Record Dates: First submitted 2019-07-11; First posted 2019-07-12 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Aging
Keywords: Very old adults; Memorizing; Motor imagery; Motor learning; Upper limb; Lower limb; Motor task; Manual task
MeSH Terms: interventions — hop protein, Drosophila

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patient aged over 80 years old will be included. They will have motor imagery training of manual task and motor imagery training of motor task.
  Interventions: Other: motor imagery as training manual task; Other: motor imagery as training motor task
- Control group (Active Comparator): Patient aged over 80 years old will be included. They will have emotionally neutral film as training of manual task and emotionally neutral film as training of motor task.
  Interventions: Other: emotionally neutral film as training of manual task; Other: emotionally neutral film as training of motor task

INTERVENTIONS:
Other: motor imagery as training manual task — They will have a motor imagery as training manual task for 30 minutes. They will have 3 tests for performing manual task before training (pretest) and after training (post-test).
  Other Names: Nine Hole Peg Test (NHPT)
  Arms: Experimental group
Other: motor imagery as training motor task — They will have a motor imagery as training motor task for 30 minutes before performing this task.
  They will have 3 tests for performing motor task before training (pretest) and after training (post-test).
  Other Names: hopscotch
  Arms: Experimental group
Other: emotionally neutral film as training of manual task — They will have to watch an emotionally neutral as training manual task for 30 minutes before performing this task.
  They will have 3 tests for performing manual task before training (pretest) and after training (post-test).
  Other Names: Nine Hole Peg Test (NHPT)
  Arms: Control group
Other: emotionally neutral film as training of motor task — They will have to watch an emotionally neutral as training motor task for 30 minutes before performing this task.
  They will have 3 tests for performing motor task before training (pretest) and after training (post-test).
  Other Names: hopscotch
  Arms: Control group

SUMMARY:
Aging is associated with impairments in cognitive function, particularly motor learning and memorizing, impacting functional capacities. Older adults are still able to learn new skills but at a slower rate, and they forget quickly the new-learned skill because of an alteration in motor memory. Motor imagery, which is a mental simulation of an action without actual execution, has been demonstrated to improve performance in young adults and stabilize performance after a short break in older adults. However, in very old adults (>80 years old) for whom the decline in motor and cognitive functions is greater, it is unknown whether motor imagery training during a short break is still efficient. Previous studies on old adults were performed on upper limb muscles. Because aging differentially affects upper and lower limb muscles, the present study will aim to explore the effects of motor imagery on motor memorizing in both upper and lower limb muscles.

DETAILED DESCRIPTION:
The primary purpose is to evaluate the effectiveness of motor imagery to improve the performance of very old people (> 80 years) through learning a task of the upper limbs.

ELIGIBILITY:
Inclusion Criteria:

* Being part of the Proof cohort
* Signed written consent form
* Affiliated to social security

Exclusion Criteria:

* Pathology or chirurgical intervention causing locomotor disorder
* Neurological or psychic pathology
* Use psychotropic drugs
* Mini-Mental State Examination (MMSE) < 20

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Performance at the manual task (Nine Hole Peg Test (NHPT)) (s) | Day: 0
  Comparison of performance at the manual task (Nine Hole Peg Test (NHPT)) results in post-test between experimental and control group. Measured in seconds when performing manual task.

SECONDARY OUTCOMES:
Performance at the motor task (s) | Day: 7
  Comparison of performance at the motor task (hopscotch) results pre-test and post-test between experimental and control group.
  Measured in number of tests.
Learning capacity of manual task (Nine Hole Peg Test (NHPT)) | Day: 0
  Comparison of manual task (Nine Hole Peg Test (NHPT)) results between pre-test and post-test.
  Measured in seconds.
Learning capacity of motor task (hopscotch) | Day: 7
  Comparison of motor task (hopscotch) results between pre-test and post-test. Measured in number of tests.
Test of 6 minutes walking (m) | Day: 0
  Comparison of test of 6 minutes walking results between experimental and control group. Measured in meters.
Test of Get-up-and-Go (s) | Day: 0
  Comparison of test of Get-up-and-Go results between experimental and control group.
  For test of Get-up-and-Go, participants will be asked to stand from a seated position, walk 3 meters at their usual pace, turn around, walk back to the chair, and sit down.
  Measured in seconds when performing test.

CONTACTS AND LOCATIONS:
Overall Officials: Léonard FEASSON, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No